CLINICAL TRIAL: NCT04610320
Title: A Phase 1 Study of Daratumumab-SC for Reduction of Circulating Antibodies in Patients With High Allosensitization Awaiting Heart Transplantation
Brief Title: Daratumumab-SC for Highly Sensitized Patients Awaiting Heart Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ronald Witteles (Other)
Responsible Party: Sponsor-Investigator, Ronald Witteles, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53476
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Allosensitization; Heart Transplant Failure and Rejection
Keywords: Immunotherapy, anti-CD38 antibody
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daratumumab-SC Injection (Experimental): * Participants will receive a subcutaneous dose of Daratumumab-SC (1800 mg) weekly for 8 doses and then every other week for 2 doses.
  * Participants will undergo laboratory testing, including for circulating antibodies, at baseline, prior to each infusion session, and at the end of the study.
  Interventions: Drug: Daratumumab-SC

INTERVENTIONS:
Drug: Daratumumab-SC — >Daratumumab-SC 1800 mg subcutaneous weekly for 8 doses and then every other week for 2 doses.

SUMMARY:
The purpose of this study is to test whether Daratumumab-SC, a drug that eliminates antibody-producing plasma cells, can effectively lower the level of preformed antibodies in patients awaiting heart transplantation. These preformed antibodies limit the number of donor hearts that are compatible for the patients. If Daratumumab-SC can effectively remove preformed, donor-specific antibodies, then highly allosensitized patients will have more compatible hearts available to them, potentially decreasing transplant waitlist time and reducing mortality.

ELIGIBILITY:
Inclusion Criteria:

* Participant is on an active list for a heart transplant.
* Participant has a high level of allosensitization, defined as a calculated PRA (panel of reactive antibodies) of 50%, based on their antibody status at the time of entry into the study.
* Ability to understand and willingness to sign an informed consent form prior to any study-related procedures.
* Women of childbearing potential must have a negative pregnancy test at screening.
* Both male and female patients must use effective methods of birth control, must not donate eggs or sperm during the course of the study and for 3 months after stopping daratumumab-SC.
* Adequate bone marrow function.
* Adequate renal function (estimated GFR greater than or equal to 15 mL/min by the Cockcroft-Gault formula).

Exclusion Criteria:

* History of allergy or intolerance to daratumumab or Daratumumab-SC.
* Prior diagnosis of myeloma or light chain amyloidosis.
* Active infection.
* Women who are pregnant or breastfeeding.
* Ongoing desensitization treatment with another agent. Subjects are excluded if they have received:

  * a. IVIG within 30 days of enrollment.
  * b. Proteasome inhibitor within 60 days of enrollment.
  * c. Rituximab within 180 days of enrollment.
* Any condition which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the Investigator, unacceptably increase the subject's risk by participating in the study.
* Contraindication to herpes zoster prophylaxis.
* Known to be seropositive for human immunodeficiency virus (HIV).
* Known to be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
* Known to be seropositive for hepatitis C (except in the setting of a sustained virologic response (SVR), defined as aviremia at least 12 weeks after completion of antiviral therapy).
* Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and subjects must be excluded if FEV1 is <50% of predicted normal.
* Known moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification.
* Known history of human immunodeficiency virus (HIV).
* History of blood product transfusion within 60 days of enrollment, or anticipated need for blood product transfusion during the course of the study.
* Moderate-severe liver dysfunction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Change in the level of preformed HLA antibodies before and after Daratumumab-SC treatment, based on the absolute difference in PRA levels before and after treatment. | Baseline and Week 12 (or the last measurement prior to heart transplantation, whichever is earlier).
  Will assess the difference in PRA percentage (defined based on those HLA antibodies which have a mean fluorescence intensity [MFI] >3000) at baseline versus Week 12.

SECONDARY OUTCOMES:
Percent MFI change for each individual preformed HLA antibody at Week 6. | Baseline and Week 6 (or the last measurement prior to heart transplantation, whichever is earlier).
  Will measure the percent change in the MFI of each circulating preformed HLA antibody from baseline to Week 6 or the time of heart transplantation (whichever is earlier).
Percent MFI change for each individual preformed HLA antibody at Week 12. | Baseline and Week 12 (or the last measurement prior to heart transplantation, whichever is earlier).
  Will measure the percent change in the MFI of each circulating preformed HLA antibody from baseline to Week 12 or the time of heart transplantation (whichever is earlier).
Percent MFI change for each individual preformed HLA antibody at Week 15. | Baseline and Week 15 (or the last measurement prior to heart transplantation, whichever is earlier).
  Will measure the percent change in the MFI of each circulating preformed HLA antibody from baseline to Week 15 or the time of heart transplantation (whichever is earlier).
Change in the level of preformed HLA antibodies before and after Daratumumab-SC treatment, based on the absolute difference in PRA levels at baseline and Week 6. | Baseline and Week 6 (or the last measurement prior to heart transplantation, whichever is earlier).
  Will assess the difference in PRA percentage (defined based on those HLA antibodies which have a mean fluorescence intensity [MFI] >3000) at baseline versus Week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Witteles, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No